CLINICAL TRIAL: NCT05482477
Title: Timing of Transcutaneous Acupoint Electrical Stimulation on Postoperative Recovery in Geriatric Patients with Gastrointestinal Tumor：a Protocol of Randomised Controlled Trial
Brief Title: Timing of Transcutaneous Acupoint Electrical Stimulation on Postoperative Recovery in Geriatric Patients with Gastrointestinal Tumor
Acronym: TEAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Subei People's Hospital of Jiangsu Province (Other)
Responsible Party: Principal Investigator, Lijuan Xi, Nurse, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lujuan Xi
Record Dates: First submitted 2022-07-24; First posted 2022-08-01 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- preoperative TEAS group (Experimental): Receive a TEAS on bilateral Neiguan (PC6) Yintang (GV29) and Zusanli (ST36) by the transcutaneous electrical stimulators to provide an altered frequency 2/100 Hz, disperse-dense waves, and adjusted intensity which was less than 10 mA, 30 min before anesthesia.
  Interventions: Other: Transcutaneous acupoint electrical stimulation
- Intraoperative TEAS group (Experimental): Receive a TEAS on bilateral Neiguan (PC6) Yintang (GV29) and Zusanli (ST36) by the transcutaneous electrical stimulators to provide an altered frequency 2/100 Hz, disperse-dense waves, and adjusted intensity which was less than 10 mA, from 30 min before anesthesia to the end of surgery
  Interventions: Other: Transcutaneous acupoint electrical stimulation
- Postoperative TEAS group (Experimental): Receive a TEAS on bilateral Neiguan (PC6) Yintang (GV29) and Zusanli (ST36) by the transcutaneous electrical stimulators to provide an altered frequency 2/100 Hz, disperse-dense waves, and adjusted intensity which was less than 10 mA, once a day, 30 minutes each time for 7 consecutive days after operation
  Interventions: Other: Transcutaneous acupoint electrical stimulation
- Pre-and post-operative TEAS group (Experimental): Receive a TEAS on bilateral Neiguan (PC6) Yintang (GV29) and Zusanli (ST36) by the transcutaneous electrical stimulators to provide an altered frequency 2/100 Hz, disperse-dense waves, and adjusted intensity which was less than 10 mA, from 1 day before operation to 7 days after operation, once a day, 30 minutes each time.
  Interventions: Other: Transcutaneous acupoint electrical stimulation
- Perioperative TEAS group (Experimental): Receive a TEAS on bilateral Neiguan (PC6) Yintang (GV29) and Zusanli (ST36) by the transcutaneous electrical stimulators to provide an altered frequency 2/100 Hz, disperse-dense waves, and adjusted intensity which was less than 10 mA, 30 min before the induction of anesthesia to the end of the surgery, 1 day before operation, and on the 1st, 2nd and 3rd days after surgery, 30 min once a day.
  Interventions: Other: Transcutaneous acupoint electrical stimulation
- Sham TEAS group (Sham Comparator): the electrodes were placed at the same time as the perioperative TEAS group, but the electronic stimulation was not applied and they were told that the TEAS treatment have no feeling
  Interventions: Other: Transcutaneous acupoint electrical stimulation
- Control group (No Intervention): receive standardised perioperative management such as preoperative health education, optimize anaesthesia scheme, intraoperative heat preservation, and reduce surgical trauma.

INTERVENTIONS:
Other: Transcutaneous acupoint electrical stimulation — Transcutaneous electrical acupoint stimulation (TEAS) is a new type of acupoint stimulation therapy that inputs low-frequency pulse current into human acupoints through electrodes pasted on the skin surface to achieve therapeutic purposes, which combined the preponderances of both acupuncture and transcutaneous electrical nerve stimulation (TENS). TEAS is non-invasive, easy to operate and acceptable to patients. Study showed that TEAS treatment can reduce the consumption of intraoperative anesthetic and improve postoperative nausea and vomiting (PONV) and postoperative recovery.
  Arms: Intraoperative TEAS group; Perioperative TEAS group; Postoperative TEAS group; Pre-and post-operative TEAS group; Sham TEAS group; preoperative TEAS group

SUMMARY:
Postoperative cognitive dysfunction(POCD). is a central nervous system complication in cancer patients with a 8.9-46.1% incidence. It is mainly manifested as impaired memory, descending information handling ability and decline or damage of attention, perception, abstract thinking, executive, language, and body movement. However, it is difficult to identify and it can last for months or years or even become a dementia state, which can severely affect patients' postoperative recovery, prolong the hospitalization time, reduce the quality of life, increase the mortality and the consumption of family and social medical resources, and intensifies the national economic and social burden.

Transcutaneous electrical acupoint stimulation (TEAS) is a new type of acupoint stimulation therapy that inputs low-frequency pulse current into human acupoints through electrodes pasted on the skin surface to achieve therapeutic purposes, which combined the preponderances of both acupuncture and transcutaneous electrical nerve stimulation (TENS). TEAS is non-invasive, easy to operate and acceptable to patients. Study showed that TEAS treatment can reduce the consumption of intraoperative anesthetic and improve postoperative nausea and vomiting (PONV) and postoperative recovery.

Also, studies have shown that TEAS treatment may improve the cognitive function of geriatric patients. Most studies have shown that TEAS treatment 10~30 minutes before operation or from entering the operating room to the end of operation can reduce the incidence of POCD in elderly patients. Some studies showed that preoperative combined with postoperative or simple postoperative TEAS treatment can significantly improve patients' postoperative cognitive function. Our previous research showed that perioperative TEAS treatment can reduce the postoperative inflammatory response and increased the postoperative cognitive function score and decrease the incidence of POCD in geriatric patients with gastrointestinal tumor. Moreover, studies showed that long-term electroacupuncture treatment is easy to cause "tolerance effect', leading to the activation of the negative feedback mechanism of the body, and reduction of the number of receptors, and the weakening of the treatment effect. So, what is the best time period for TEAS to improve POCD and reduce the use of resources? Therefore, the objective of this study is to discuss different time of TEAS on POCD in geriatric patients with gastrointestinal tumor.

DETAILED DESCRIPTION:
Therefore, the objective of this study is to discuss different time of TEAS on POCD in geriatric patients with gastrointestinal tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years or older.

  * Patients diagnosed with gastrointestinal tumor and received radical resection of gastrointestinal tumors under general anesthesia in Subei People's Hospital of Jiangsu province.

    * Patients willing and able to give informed consent and comply with this study protocol.

      * American Society of Anesthesiology (ASA) classification I～III. ⑤ Preoperative Tilburg frailty scale score is less than 5 points. ⑥ Preoperative D-dimer was normal.

Exclusion Criteria:

* Preoperative cognitive dysfunction or history of cognitive dysfunction, dementia, and delirium.

  * History of severe depression, schizophrenia, or other mental and nervous system diseases or taking antipsychotic or antidepressant drugs in the past.

    * Patients with severe hearing or visual impairment without assistive tools.

      * Patients who have difficulty in communicating.

        * Male patients average daily pure alcohol intake ≥ 61 g or female patients average daily pure alcohol intake ≥ 41 g.

          * Patients received surgical treatment within 3 months or preoperative hospitalized over 3 months.

            * Patients with severe heart, liver, or renal failure.

              ⑧ Patients with hypoxemia (blood oxygen saturation < 94%) more than 10 min during the operation.

              ⑨ Patients admitted to ICU after operation.

              ⑩ Patients who quit or died due to noncooperation or sudden situation.

              ⑪ Patients who already participate in other clinical studies which may influence this study.

              ⑫ Patients who underwent emergency surgery.

              ⑬ Patients who had a history of acupuncture treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination(MMSE) | From preoperative to 3 days after operation
  Assess the cognitive function of the patient. The MMSE is a 30 points questionnaire used to measure orientation (time and place), memory (immediate and short term), attention, calculation, and language (naming, repetition, listening, reading, and writing) . Higher score means better cognitive function.
Auditory Verbal Learning Test-HuaShan version(AVLT-H) | From preoperative to 3 days after operation
  Assess the cognitive function of the patient. AVLT-H was used to evaluate the memory of the subjects.The subjects learned and recalled 12 words and repeated themself three times. After the nonverbal test interval of about 5min and 20min, the fourth (short delayed recall) and fifth (long delayed recall) repeat will be recorded respectively. The sixth recall was reconfirmation, that is, the data collectors read 24 words, and the subjects answered whether they had learned them. According to the knowledge level and cooperation degree of local elderly subjects, the fourth repeat will be recorded and a correct word will get 1 point.
Digital Symbol Coding(DSC) | From preoperative to 3 days after operation
  Assess the cognitive function of the patient. DSC was used to evaluate the executive function of the subjects. For the test, the subjects need to fill in the numbers corresponding to the symbols within 90s. A correct number will get 1 point, up to 90 points.
Verbal Fluency Test(VFT) | From preoperative to 3 days after operation
  Assess the cognitive function of the patient. VFT was used to evaluate the language ability of the subjects. The subjects should say as many names of animals, fruits and vegetables as possible within 1 minute. A correct object will get 1 point, no point will be given if repeated.
Clock Drawing Task(CDT) | From preoperative to 3 days after operation
  Assess the cognitive function of the patient. CDT was used to evaluate the visual spatial structure ability of the subjects. The subjects need to draw the dial of the clock on paper and write the numbers in the correct position. Scoring method: ① Draw a closed circular outline, 1 point. ②The number display and sequence in the dial are correct, 2 points. ③The position of the hour and minute hand is correct, 1 point. To reduce the learning effect, the test time preoperative and postoperative in this study is drawn at 08:10 and 07:50 respectively.

SECONDARY OUTCOMES:
Interleukin-6(IL-6) | Baseline and on the 3rd day after the operation
  Evaluate patients' postoperative inflammatory status. IL-6 is a pro-inflammatory cytokine which can mediate inflammatory and immune responses in the CNS.
S100 calcium proteinβ(S100β) | Baseline and on the 3rd day after the operation
  Evaluate patients' postoperative inflammatory status. S100β is a biomarker which existed in the cell of peripheral and central nervous system(CNS) and it may participate in the mechanism of cognitive impairment.
insulin-like growth factor-1( IGF-1 ) | Baseline and on the 3rd day after the operation
  Evaluate patients' postoperative inflammatory status. As one of the neurotrophic factors, IGF-1 has been proved to have neuroprotective and neuroproliferative effects and it may delay the degeneration of dopaminergic neurons, protect dopaminergic neurons and promote nerve regeneration through a variety of ways, including inhibiting inflammatory reaction. IGF-1 plays an important role in the survival and differentiation of neurons, and is related to a variety of neurodegenerative diseases. Studies showed that the level of serum IGF-1 in patients with Parkinson's disease(PD) is related to cognitive dysfunction, and serum IGF-1 may be a biomarker of cognitive dysfunction in patients with PD.
C-reactive protein(CRP) | Baseline and on the 3rd day after the operation
  Evaluate patients' postoperative inflammatory status. CRP is a non-specific biomarker inflammation which has been proved to accelerate the development of neurodegenerative disorders by activating microglia, increasing levels of proinflammatory cytokines, and activating the complement cascade.
Numerical pain score(NRS) | on the third day after operation
  Evaluate the postoperative recovery of patients. On the scale of the 10 point system, the self rating is based on the degree, which is divided into 1-10 levels. According to the corresponding numbers, the pain can be divided into different degrees, that is, level 0 means no pain, level 1-3 means mild pain, level 4-6 means moderate pain, and level 7-10 means severe pain.
Score of Branden pressure ulcer risk assessment scale(Branden) | The seventh day after operation
  Branden is divided into six dimensions: perception, humidity, activity mode, activity ability, nutrition, friction and shear force. The friction and shear force are rated at Level 3, and the rest are rated at level 4, with a score range of 6-23 points. The higher the score, the smaller the risk of pressure ulcer occurrence, with 15-18 points for mild risk, 13-14 points for moderate risk, 10-12 points for high risk, and ≤ 9 points for serious risk.
Score of Barthel index (BI) | The seventh day after operation
  BI is a tool widely used in clinic to evaluate patients'activities of daily living(ADL). It includes 10 items, including diet, bed and wheelchair transfer, personal hygiene, toileting, bathing, walking, going up and down stairs, dressing, defecation control and urination control, with a total score of 100 points. If the score is in the range of 0 ~ 40 points, it belongs to severe ADL deficiency; if it is in the range of 41 ~ 60 points, it belongs to moderate ADL deficiency; if it is in the range of 61 ~ 100 points, it belongs to mild ADL deficiency. The BI scale can be evaluated by asking patients or their families, which is simple, fast and highly reliability.
Telephone Interview for Cognitive Status-Modified(TICS-m) | 1, 3, 6 months after operation.
  Assess the cognitive function of the patient. TICS-m is modified from the earliest version of TICS which is modeled on MMSE. Gallo and Breitiner revised the original version, adding tests such as delayed memory of words and five times of phone tapping, and expanded it to 21 items, with a total score of 50 points. It can be divided into three parts: memory (20 points), orientation (13 points), language and attention (17 points). The higher the score, the better the condition of the project. <28 points is defined as dementia, 28~32 points is defined as mild cognitive impairment(MCI). More over the TICS-m has been proved to have good reliability and validity in the Chinese population.
Postoperative exhaust time | The second day after operation
  Record the first anal exhaust time after operation
Postoperative defecation time | The second day after operation
  Record the first defecation time after operation
Postoperative eating time | The second day after operation
  Record the first eating time after operation
The time of get out of bed for the first time after operation | The second day after operation
  Record the time of get out of bed for the first time after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin X, Chen Y, Zhang P, Chen G, Zhou Y, Yu X. The potential mechanism of postoperative cognitive dysfunction in older people. Exp Gerontol. 2020 Feb;130:110791. doi: 10.1016/j.exger.2019.110791. Epub 2019 Nov 23. PMID 31765741
- [Background] Deiner S, Liu X, Lin HM, Jacoby R, Kim J, Baxter MG, Sieber F, Boockvar K, Sano M. Does Postoperative Cognitive Decline Result in New Disability After Surgery? Ann Surg. 2021 Dec 1;274(6):e1108-e1114. doi: 10.1097/SLA.0000000000003764. PMID 32149824
- [Background] Liu J, Huang K, Zhu B, Zhou B, Ahmad Harb AK, Liu L, Wu X. Neuropsychological Tests in Post-operative Cognitive Dysfunction: Methods and Applications. Front Psychol. 2021 Jun 4;12:684307. doi: 10.3389/fpsyg.2021.684307. eCollection 2021. PMID 34149572
- [Background] Xi L, Fang F, Yuan H, Wang D. Transcutaneous electrical acupoint stimulation for postoperative cognitive dysfunction in geriatric patients with gastrointestinal tumor: a randomized controlled trial. Trials. 2021 Aug 23;22(1):563. doi: 10.1186/s13063-021-05534-9. PMID 34425851
- [Background] Ricci M, Graef S, Blundo C, Miller LA. Using the Rey Auditory Verbal Learning Test (RAVLT) to differentiate alzheimer's dementia and behavioural variant fronto-temporal dementia. Clin Neuropsychol. 2012;26(6):926-41. doi: 10.1080/13854046.2012.704073. Epub 2012 Jul 18. PMID 22809061
- [Background] Wessels AM, Lines C, Stern RA, Kost J, Voss T, Mozley LH, Furtek C, Mukai Y, Aisen PS, Cummings JL, Tariot PN, Vellas B, Dupre N, Randolph C, Michelson D, Andersen SW, Shering C, Sims JR, Egan MF. Cognitive outcomes in trials of two BACE inhibitors in Alzheimer's disease. Alzheimers Dement. 2020 Nov;16(11):1483-1492. doi: 10.1002/alz.12164. Epub 2020 Oct 13. PMID 33049114
- [Background] Bertola L, Mota NB, Copelli M, Rivero T, Diniz BS, Romano-Silva MA, Ribeiro S, Malloy-Diniz LF. Graph analysis of verbal fluency test discriminate between patients with Alzheimer's disease, mild cognitive impairment and normal elderly controls. Front Aging Neurosci. 2014 Jul 29;6:185. doi: 10.3389/fnagi.2014.00185. eCollection 2014. PMID 25120480
- [Background] Leissing-Desprez C, Thomas E, Segaux L, Broussier A, Oubaya N, Marie-Nelly N, Laurent M, Cleret de Langavant L, Fromentin I, David JP, Bastuji-Garin S. Understated Cognitive Impairment Assessed with the Clock-Drawing Test in Community-Dwelling Individuals Aged >/=50 Years. J Am Med Dir Assoc. 2020 Nov;21(11):1658-1664. doi: 10.1016/j.jamda.2020.03.016. Epub 2020 May 6. PMID 32387111
- [Derived] Yin W, Fang F, Zhang Y, Xi L. Timing of transcutaneous acupoint electrical stimulation for postoperative recovery in geriatric patients with gastrointestinal tumors: study protocol for a randomized controlled trial. Front Med (Lausanne). 2025 Mar 5;12:1497647. doi: 10.3389/fmed.2025.1497647. eCollection 2025. PMID 40109717